CLINICAL TRIAL: NCT01879813
Title: A Randomised, Double-blind, Parallel Groups, Placebo-controlled 6 Weeks Human Intervention Study Investigating the Effect of a Phospholipid Drink on Cognitive Performance
Brief Title: The Effect of a Phospholipid Drink on Cognitive Performance Under Acute Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Principal Investigator, Prof Louise Dye, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Stress and cognition study
Record Dates: First submitted 2012-10-15; First posted 2013-06-18 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Cognitive Performance (Focus)
Keywords: Memory; Attention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phospholipid drink (Active Comparator): Participants will consume a phospholipid drink daily for 6 weeks
  Interventions: Dietary Supplement: Phospholipid drink
- Placebo milk drink (Placebo Comparator): Participants will consume a placebo drink (no added phospholipids) daily for 6 weeks
  Interventions: Dietary Supplement: Placebo milk drink

INTERVENTIONS:
Dietary Supplement: Phospholipid drink — Participant in an intervention parallel group will consume a drink with added phospholipids
  Arms: Phospholipid drink
Dietary Supplement: Placebo milk drink — Participant in an intervention parallel group will consume a drink without added phospholipids
  Arms: Placebo milk drink

SUMMARY:
The study will explore the effects of a 6-week phospholipid drink intervention on the cognitive performance and physiological and subjective stress parameters of males following a repeated psychosocial/physical stressor.

DETAILED DESCRIPTION:
The study conforms to a randomised, double-blind, placebo controlled, parallel groups design examining cognitive performance and physiological/subjective stress responses after a psychosocial/physical stressor before and after a six week daily intake of an phospholipid containing drink vs. placebo.

The study will examine:

Cognitive performance following acute stress prior to, and following 6-weeks intake of a phospholipid containing drink or a placebo analogue.

Physiological and subjective stress responses following acute stress prior to, and following 6-weeks intake of a phospholipid containing drink or a placebo analogue

ELIGIBILITY:
Inclusion Criteria:

* Male ≥18 years old
* Healthy (self-report health questionnaire)
* BMI <30 kg/m²
* Free from medication (prescribed and 'over-the-counter')

Exclusion Criteria:

* Current psychological affective/mood disorders
* Self-reported physical disorder/disease (significant cardiovascular, autoimmune, endocrine, gastrointestinal or neurological conditions, chronic pain, or sleep disorders)
* High chronic stress
* Smokers
* Recreational drug use (within the last month)
* Night shift work
* Hypertension (resting blood pressure exceeding 160/95 mmHg)
* Skin conditions (e.g. eczema) on hands
* Food allergies
* Participation in a clinical study within a month prior to screening or during participation
* Participation in any of our previous stress induction studies

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cognitive performance change from baseline | Week 1 (baseline) and week 6
  Performance on a cognitive test battery at baseline will be compared to performance at week 6

SECONDARY OUTCOMES:
Salivary cortisol change from baseline | Week 1 (baseline) and week 6
  Salivettes will be used to collect salivary cortisol response across exposure to a laboratory stress protocol on two occasions separated by 6 weeks
Blood pressure (systolic/diastolic) change from baseline | Week 1 (baseline) and week 6
  An ambulatory blood pressure monitor will be used to collect blood pressure response profiles across exposure to a laboratory stress protocol on two occasions separated by 6 weeks
Heart rate change from baseline | Week 1 (baseline) and 6 weeks
  An ambulatory blood pressure monitor will be used to collect heart rate response profiles across exposure to a laboratory stress protocol on two occasions separated by 6 weeks
Subjective stress change from baseline | Week 1 (baseline) and 6 weeks
  The Stress and Arousal Checklist (Mackay, 1978)will be used to collect subjective stress response profiles across exposure to a laboratory stress protocol on two occasions separated by 6 weeks
Subjective mood change from baseline | Week 1 (baseline) and 6 weeks
  The Profile of Mood States (Mc Nair et al., 1971)will be used to collect subjective mood response profiles across exposure to a laboratory stress protocol on two occasions separated by 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Louise Dye, PhD, Principal Investigator — University of Leeds
Locations (1):
- Human Appetite Research Unit, University of Leeds, Leeds, West Yorkshire, United Kingdom